CLINICAL TRIAL: NCT04584138
Title: Eye Movement During Autobiographical Memory in Alzheimer's Disease
Brief Title: Autobiographical Memory
Acronym: EMAM
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0322
Record Dates: First submitted 2020-09-23; First posted 2020-10-12 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer's Disease; Autobiographical Memory; Eye Movement; Memory
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Study of eye movements — The assessment of eye movement during autobiographical retrieval (i.e., retrieval of personal memories) in patients with Alzheimer's Disease.

SUMMARY:
This study aims at the assessment of eye movement during autobiographical retrieval (i.e., retrieval of personal memories) in patients with Alzheimer's Disease.

DETAILED DESCRIPTION:
There is an increased interest in the study of eye movements during the retrieval of autobiographical memories and recent research has demonstrated how retrieval of autobiographical memory can activate eye movement. This research has been however mainly concerned with young adults and, until now, little is known about the relationship between eye movement and autobiographical memory in patients with Alzheimer's Disease. The aim of the current study is therefore to evaluate eye movements during the retrieval of autobiographical memories in patients with Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria :

* Diagnosis of Alzheimer's Disease at the mild stage

Exclusion Criteria :

* Neurological/psychiatric disorders (other than Alzheimer's Disease)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Alzheimer's disease in the mild stage
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Number of fixations and saccades | Four weeks (from assessment till analysis)
  Number
Duration of fixations and saccades | Four weeks (from assessment till analysis)
  Duration in milliseconds

SECONDARY OUTCOMES:
Pupil size | Four weeks (from assessment till analysis)
  In millimeter

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] El Haj M, M J Janssen S, Gallouj K, Lenoble Q. Autobiographical Memory Increases Pupil Dilation. Transl Neurosci. 2019 Dec 19;10:280-287. doi: 10.1515/tnsci-2019-0044. eCollection 2019. PMID 31915538
- See also: Autobiographical Memory Increases Pupil Dilation — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6943370/